CLINICAL TRIAL: NCT04932746
Title: The Effect of Dexmedetomidine on Oxygen and Intrapulmonary Shunt During One Lung Ventilation in Pediatric Surgery: Randomized Controlled Trial
Brief Title: The Effect of Dexmedetomidine on Oxygen During One Lung Ventilation in Pediatric Surgery.
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: University Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UDMS-Anesth-01-2021
Record Dates: First submitted 2021-05-23; First posted 2021-06-21 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: One Lung Ventilation OLV; Esophageal Atresia; Hydrocystoma; Pneumonectomy; Pleura; Abscess
Keywords: Dexmedetomidine; One lung ventilation OLV; Hypoxic pulmonary vasoconstriction HPV; Pulmonary shunt fraction Qs / Qt
MeSH Terms: conditions — Esophageal Atresia; Hidrocystoma; Abscess | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple masking:
  Anesthesiologists, graduate students, anesthesiologists, patients and their families will not know if a child is taking the drug or not.
  Also, the person who will conduct the survey will not know either, all will be hidden.
  Depending on the volume in ml, to mask the medical team from the substance of the drug...
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The dexmedetomidine group: (Experimental): An initial dose of 1 mcg / kg 1 dexmedetomidine will be given 10 minutes after the start of anesthesia infusion within 10 minutes, after which the dexmedetomidine infusion is maintained at a dose of 0.4 mcg / kg / hour.
  The injection will be stopped before the skin is closed.
  Interventions: Drug: Dexmedetomidine
- The Placebo group (the control group): (Experimental): After the same anesthesia, the same amount of Saline solution will be administered, instead of dexmedetomidine, with the same protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Infusion syringes are supplied with a concentration of 0.25 mcg / mL (dexmedetomidine or placebo) either 80 mcg / 20 mL, 200 mcg / 50 mL, or 400 mcg / 100 mL.
  It begins with infusion of 4 ml within 10 minutes and then continues infusion, depending on the child's weight, at 1.6 ml / kg / h.
  All injections will be prepared randomly by a doctor who did not participate in the study, and then placed in unmarked infusion pumps, given to an anesthesiologist (more than 10 years experience in pediatric anesthesia) without knowledge of the infusion content. The randomization process is carried out via sealed envelope technique.
  The injections in both groups will be stopped before the skin is closed. Both patients and anesthesiologists blinded the study drug (dexmedetomidine or placebo) by infusion of solution (dexmedetomidine or placebo). Depending on the size in ml, to ensure that there is no bias and blindness to the medical team about what the drug is.
  Other Names: Precedex
  Arms: The dexmedetomidine group:
Drug: Placebo — The same anesthesia, the same amount of Saline solution will be administered, instead of dexmedetomidine, with the same protocol
  Other Names: Saline
  Arms: The Placebo group (the control group):

SUMMARY:
The children who will undergo OLV (one lung ventilation) through general anesthesia will be divided into two groups:

The first will be intravenous infusion of dexmedetomidine at 0.4 mcg / kg / hour, and the second will be intravenous infusion of normal saline.

We will take three samples of arterial blood gas (ABG) during the surgery at certain times. We record the hemodynamic values, PaO2, and calculate the value of the shunt Qs / Qt.

DETAILED DESCRIPTION:
Lung isolation or one lung ventilation OLV means the mechanical separation of the lungs with independent ventilation of one lung from the other, in order to provide a suitable space for the work of the surgeon, and to protect a healthy lung from bleeding or edema caused by lung damage. OLV can lead to a mismatch in the ventilation / perfusion (V / Q) ratio resulting in increased intrapulmonary shunt as well as hypoxia.

Hypoxic pulmonary vasoconstriction HPV is the most important preventive mechanism against hypoxemia, as blood flow moves from the unventilated lung to the ventilated lung to maintain an adequate arterial oxygen transport rate, HPV is a defense mechanism against hypoxia as it reduces pulmonary shunt. So that there is less oxygen drop than expected. HPV reaches its maximum effect in 15 minutes, resulting in decreased pulmonary shunt, homogenization of ventilation / perfusion ratio, and improved oxygen delivery. HPV is affected by various factors: changes in pulmonary pressure, alkalosis, vasodilators, anesthetic agents etc. Among these factors, anesthetic inhaled gases have the greatest effect on HPV.

Pulmonary shunt: It is the sum of the physiological shunt (poorly ventilated air sacs) and the anatomical shunt and the pulmonary shunt fraction (Qs/Qt) is calculated from the equation Qs/Qt = (CcO2 - CaO2)/(CcO2 - CvO2) Qs: blood flow through the shunt, Qt : total blood flow, Cc'O2 : pulmonary capillary content of O2, CaO2 : arterial content of O2, CvO2 : venous mixed content of O2 100% O2 test: often performed in a cardiac catheterization lab, operating room, or ICU, the patient breathes 100% O2 until nitrogen is washed out from their lungs (20 minutes). The oxygen concentration even in poorly ventilated units will approach 100%. This means that the partial pressure and blood saturation are equal in the poorly ventilated and well-ventilated alveolar units, thus the physiological pulmonary shunt is canceled and the anatomical pulmonary shunt remains After lung isolation and OLV application, we perform anesthesia maneuvers on the ventilator and adjust the applied ventilators in order to maintain adequate oxygenation of the patient: increased PEEP, increased FLOW, increased tidal volume Vt, increased Pmax, increased FiO2, thus eliminating the physiological pulmonary shunt and the anatomical pulmonary shunt remains, in total we apply 100% O2 testing.

Dexmedetomidine is a selective agonist for α2 receptors whose affinity for α2 receptors is eight times more than clonidine. At a dose of 0.3 mg / kg it activates protein G and inhibits norepinephrine secretion. When given in larger doses or infusion it stimulates the peripheral α2 receptors; It reduces the levels of norepinephrine in the plasma by more than 90%, thus reducing the cells' metabolism and their need for oxygen.Sympathetic blocker: Reduces heart rate, blood pressure and oxygen consumption of the heart muscle. Studies have shown that alpha-adrenergic blockade abolished pulmonary vasoconstriction that responds to norepinephrine but not to hypoxia. That is, it does not affect the blood supply and HPV of the unventilated lung, widens the blood vessels of the ventilated lung, and reduces the anesthetic requirements (affecting HPV); Reduces 30% of the need for propofol; It reduces desflurane concentration and its subsequent inhibitory effect on HPV. It may also lead to transient increases in pulmonary artery pressure related to its direct effects on vascular smooth muscle through alpha-adrenergic receptors.

ELIGIBILITY:
Inclusion Criteria:

1. As per the American Society of Anesthesiologists (ASA) classification I-I physical condition children undergoing thoracic surgery with OLV.
2. From one day old to 12 years old.
3. There is no prejudice in terms of gender.
4. This study practically does not exclude any child who will undergo OLV even in the presence of cardiac, renal or hepatic diseases.

Or even in the presence of cardiac stimulants and supports (dopamine or dopamine), provided that the general condition is stable, which allows surgery and OLV.

Exclusion Criteria:

1. Premature infants: due to immaturity of the lung and insufficient formation of the surfactant.
2. Cystic Fibrosis: The depressor for surfactant and lung immaturity is not permitted to perform the OLV technique
3. There is no contraindication for the administration of dexmedetomidine in children except those who show signs of allergy to the dexmedetomidine.
4. This study does not exclude practically any child who will undergo OLV.
5. During operating surgery: The child is excluded from the study if hypoxia occurs (SpO2 <90%) and did not respond to maneuvers and anesthetic techniques (Increase PEEP Increase the FLOW, Tidal volume, increase Vt, Pmax increased pressure, FiO2 increased) Then the lungs are periodically ventilated with positive pressure, and the OLV technique is switched off and the child is excluded from the pilot study.
6. During operating surgery: If there is a drop-in heart rate less than 60 beats / minute and it does not respond to atropine or an increased dose of Cardiac tonics (dopamine).

At this time the infusion of dexmedetomidine is stopped, it is assumed that there is no very slow pulse, and if it does, it is likely that the primary cardiac lesion is the cause.

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in PaO2 during surgery | Three measurements will be taken over three times: T1: 10 min after induction of anesthesia and before OLV, T2: 10 min after lung isolation and OLV single lung ventilation, and T3: 60 min after OLV procedure.
  PaO2 : The partial pressure of oxygen The partial pressure of oxygen, also known as PaO2, is a measurement of oxygen pressure in arterial blood. It reflects how well oxygen is able to move from the lungs to the blood
Evaluation of change in Qs/Qt during surgery. Qs/Qt: is a measurement of pulmonary shunt. Qs: blood flow through the shunt, Qt : total blood flow. | Three measurements will be taken over three times: T1: 10 min after induction of anesthesia and before OLV, T2: 10 min after lung isolation and OLV single lung ventilation, and T3: 60 min after OLV procedure.
  It describes the percentage of blood that reaches the left side of the heart without picking up oxygen. The pulmonary shunt fraction (Qs/Qt) is calculated from the equation Qs/Qt = (CcO2 - CaO2)/(CcO2 - CvO2)
  Parameters we need to the equation:
  1. Measurement of arterial blood gases ABG from arteries (radial or aorta) and the values it provides:
     1. PaO2: partial pressure of arterial oxygen
     2. SaO2: the degree of oxygen saturation of arterial hemoglobin
     3. Hb: hemoglobin
  2. Measurement of ABG from the pulmonary artery or from the right atrium via central catheter
     1. PvO2: partial pressure of venous oxygen
     2. SvO2: the degree of oxygen saturation of venous hemoglobin
     3. Hb: hemoglobin
  3. The following values
     1. PB = (759 ~ 760) atmospheric pressure
     2. PH2O = 47 water vapor pressure at a body temperature of 37
     3. RQ = 0.8: RER = respiratory exchange rate when anesthetized
     4. FiO2 The Fraction of Inspired Oxygen

SECONDARY OUTCOMES:
Evaluation of change in CaO2 during surgery | Three measurements will be taken over three times: T1: 10 min after induction of anesthesia and before OLV, T2: 10 min after lung isolation and OLV single lung ventilation, and T3: 60 min after OLV procedure.
  CaO2 :arterial content of O2. CaO2 = (PaO2 × 0.0031) + (Hb × 1.36 × SaO2)
Evaluation of change in CvO2 during surgery | Three measurements will be taken over three times: T1: 10 min after induction of anesthesia and before OLV, T2: 10 min after lung isolation and OLV single lung ventilation, and T3: 60 min after OLV procedure.
  CvO2 :venous mixed content of O2. CvO2 = (PvO2 × 0.0031) + (Hb × 1.36 × SvO2)
Evaluation of change in Cc'O2 during surgery | Three measurements will be taken over three times: T1: 10 min after induction of anesthesia and before OLV, T2: 10 min after lung isolation and OLV single lung ventilation, and T3: 60 min after OLV procedure.
  Cc'O2 : pulmonary capillary content of O2. CcO2 = ([FiO2 × (PB -PH2o) - PaCO2/RQ] × 0.0031) + (Hb × 1.36)

CONTACTS AND LOCATIONS:
Overall Officials: Faten Rostom, PHD, Study Chair — Head of the Department of Anesthesiology Al-Assad University Hospital
Locations (1):
- University Children's Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asri S, Hosseinzadeh H, Eydi M, Marahem M, Dehghani A, Soleimanpour H. Effect of Dexmedetomidine Combined with Inhalation of Isoflurane on Oxygenation Following One-Lung Ventilation in Thoracic Surgery. Anesth Pain Med. 2020 Feb 12;10(1):e95287. doi: 10.5812/aapm.95287. eCollection 2020 Feb. PMID 32309196
- [Background] Huang SQ, Zhang J, Zhang XX, Liu L, Yu Y, Kang XH, Wu XM, Zhu SM. Can Dexmedetomidine Improve Arterial Oxygenation and Intrapulmonary Shunt during One-lung Ventilation in Adults Undergoing Thoracic Surgery? A Meta-analysis of Randomized, Placebo-controlled Trials. Chin Med J (Engl). 2017 Jul 20;130(14):1707-1714. doi: 10.4103/0366-6999.209891. PMID 28685722
- [Background] Lin J, Li JB, Lu Z. Clinical application and effect of dexmedetomidine in combination with continuous positive airway pressure on one-lung ventilation in lung surgery of elder patients. Pak J Pharm Sci. 2018 Nov;31(6(Special)):2879-2883. PMID 30630803
- [Background] Meng J, Lv Q, Yao J, Wang S, Yang K. Effect of Dexmedetomidine on Postoperative Lung Injury during One-Lung Ventilation in Thoracoscopic Surgery. Biomed Res Int. 2020 Oct 5;2020:4976205. doi: 10.1155/2020/4976205. eCollection 2020. PMID 33083468
- [Background] Shen Q, Xu G, Liu J, Wang L, Zhou Y, Yu Y, Lv C, Liu X. Dexmedetomidine alleviates non-ventilation associated lung injury via modulating immunology phenotypes of macrophages. Life Sci. 2020 Oct 15;259:118249. doi: 10.1016/j.lfs.2020.118249. Epub 2020 Aug 13. PMID 32798558
- [Background] Sheybani S, Attar AS, Golshan S, Sheibani S, Rajabian M. Effect of propofol and isoflurane on gas exchange parameters following one-lung ventilation in thoracic surgery: a double-blinded randomized controlled clinical trial. Electron Physician. 2018 Feb 25;10(2):6346-6353. doi: 10.19082/6346. eCollection 2018 Feb. PMID 29629058
- [Background] Wang J, Yi X, Jiang L, Dong H, Feng W, Wang S, Chu C. Protective effects of dexmedetomidine on lung in rats with one-lung ventilation. Exp Ther Med. 2019 Jan;17(1):187-192. doi: 10.3892/etm.2018.6952. Epub 2018 Nov 9. PMID 30651781
- [Background] Xie Y, Jiang W, Zhao L, Wu Y, Xie H. Effect of dexmedetomidine on perioperative inflammation and lung protection in elderly patients undergoing radical resection of lung cancer. Int J Clin Exp Pathol. 2020 Oct 1;13(10):2544-2553. eCollection 2020. PMID 33165407
- [Background] Xu B, Gao H, Li D, Hu C, Yang J. Nebulized dexmedetomidine improves pulmonary shunt and lung mechanics during one-lung ventilation: a randomized clinical controlled trial. PeerJ. 2020 Jun 5;8:e9247. doi: 10.7717/peerj.9247. eCollection 2020. PMID 32547872